CLINICAL TRIAL: NCT05574881
Title: A Prospective, Single Center, Phase II Trial of Dalpiciclib, Fulvestrant, Trastuzumab and Pertuzumab in HR Positive, HER2 Positive Metastatic Breast Cancer
Brief Title: Dalpiciclib, Fulvestrant, Trastuzumab and Pertuzumab in HR Positive, HER2 Positive Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOUNGBC-22
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: HR positive, HER2 positive Metastatic Breast Cancer; Dalpiciclib, Fulvestrant, Trastuzumab and Pertuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Fulvestrant; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): Dalpiciclib 150 mg qd; Fulvestrant 500mg d1, 15, 29, and then q4w; Pertuzumab 840mg q3w, and then 420 mg q3w; Trastuzumab 8 mg/kg q3w, and then 6 mg/kg q3w
  Interventions: Drug: Dalpiciclib; Drug: Fulvestrant; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Dalpiciclib — 150 mg qd
Drug: Fulvestrant — 500mg d1, 15, 29, and then q4w
Drug: Pertuzumab — 840mg q3w, and then 420 mg q3w
Drug: Trastuzumab — 8 mg/kg q3w, and then 6 mg/kg q3w

SUMMARY:
To investigate the efficacy and safety of Dalpiciclib, Fulvestrant, Trastuzumab and Pertuzumab in HR+/HER2+ Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily joined the study, signed informed consent, and had good compliance.
2. Postmenopausal or premenopausal perimenopausal female patients aged ≥ 18 years, Meet one of the following:

   Previous bilateral oophorectomy, or age ≥ 60 years; or Age <60, natural postmenopausal state (defined as regular months for at least 12 consecutive months After spontaneous cessation and no other pathological or physiological reasons), E2 and follicle stimulating hormone (FSH) in menopause Post-level; or Pre-menopausal or perimenopausal female patients can also be included, but must be willing to receive treatment with luteinizing hormone releasing hormone (LHRH) agonists;
3. Patients with HR+/HER2+ recurrent or metastatic breast cancer confirmed by histopathology； HER2 positivity is defined by standard of 3+ staining by immunohistochemical staining (IHC) or positive for in situ hybridization (ISH)； Estrogen receptor (ER) or Progesterone receptor (PR) positive is defined as the percentage of cells positive for ER or PR expression ≥ 10%； Local recurrence needs to be confirmed by the physician that is unresectable
4. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
5. No systemic treatment in metastatic setting. At least 12-month interval between the time of last dose of trastuzumab in adjuvant treatment and the date of diagnosis with recurrent or metastatic breast cancer
6. Had received endocrine therapy in adjuvant setting.
7. Eastern Cooperative Oncology Group Performance Status of 0-1.
8. Life expectancy ≥ 12 weeks.
9. Adequate function of major organs meets the following requirements (no blood components and cell growth factors have been used within 14 days before randomization):

Neutrophils ≥ 1.5×10^9/L， Platelets ≥ 100×10^9/L， Hemoglobin ≥ 90g/L， Total bilirubin≤ 1.5 × the upper limit of normal (ULN)， Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN， blood urea nitrogen(BUN) and Cr ≤ 1.5 × ULN， Left ventricular ejection fraction (LVEF) ≥ 50%， QTcF(Fridericia correction) ≤ 470 ms， International normalized ratio(INR)≤1.5 × ULN， activated partial thromboplastin time(APTT) ≤ 1.5 × ULN

Exclusion Criteria:

1. Meningeal metastasis or active brain parenchymal metastasis. Patients with clinically stable brain parenchymal metastases can be included, including asymptomatic brain metastases that have not received local treatment; or patients who have previously received central nervous system metastasis therapy (radiotherapy or surgery), if imaging confirms that stability has been maintained for at least 4 weeks, and have stopped symptomatic treatment (including hormones and mannitol, etc.) for more than 2 weeks
2. Visceral crisis.
3. Previously received any CDK4/6 inhibitor treatment.
4. Inability to swallow, intestinal obstruction or other factors affecting the administration and absorption of the drug.
5. Patients with other malignant tumors within 5 years or at the same time( except for cured skin basal cell carcinoma and cervical carcinoma in situ).
6. Have undergone major surgical procedures or significant trauma within 4 weeks prior to randomization, or are expected to undergo major surgery.
7. Pregnant women, lactating female, or women of childbearing age who are unwilling to take effective contraceptive measures.
8. Have a history of allergies to the drug components of this regimen.
9. Patients with active HBV and HCV infection; stable hepatitis B after drug treatment (HBV virus copy number is higher than the upper limit of reference value) and cured hepatitis C patients (HCV virus copy number exceeds the lower limit of detection method).
10. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation.
11. History of cardiac dysfunction, include (1)angina (2)clinical significant arrythmia or require drug intervention (3)myocardial infarction (4)heart failure (5) other cardiac dysfunction (judged by the physician); any cardiac or nephric abnormal ≥ grade 2 found in screening.
12. Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
13. Childbearing female who refuses to accept any contraception practice.
14. Determined by the physician, any serious coexisting disease might be harmful to the patient's safety or avoid the patients from accomplishing the treatment(e.g serious hypertension, diabetes, thyroid dysfunction,active infection etc.).
15. History of neurological or psychiatric disorders, including epilepsy or dementia.
16. Severe infections within 4 weeks prior to first dose (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs according to clinical protocols), or unexplained fever (T > 38.3 °C ) during screening or prior to first administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 6 weeks
  Safety
Objective response rate (ORR) | 6 weeks
  Proportion of subjects whose efficacy was evaluated as Complete Response(CR)/PR
Clinical benefit rate (CBR) | 6 weeks
  Proportion of subjects with CR, PR and SD≥24 weeks during the study
Duration of remission (DoR) | 6 weeks
  The time from the first assessment of CR or PR to the first assessment of Progressive Disease(PD) or death from any cause；
Overall Survival (OS) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China